CLINICAL TRIAL: NCT01855945
Title: Phase I Multi-center, Observer-Blind, Randomized, Dose-Ranging Study of Adjuvanted and Non-Adjuvanted Cell Culture-Derived, Inactivated Novel Swine Origin A/H3N2v Monovalent Subunit Influenza Virus Vaccine (H3N2c) in Children Ages 3 to <9 Years, Adolescents 9 to <18 Years, Adults 18 to < 65 Years and Elderly ≥ 65 Years and Older.
Brief Title: Safety and Immunogenicity of Three Dosage Levels of Swine Influenza Vaccine in Children Ages 3 to <9 Years, Adolescents 9 to <18 Years, Adults 18 to <65 Years and Elderly 65 Years and Older.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V129_01
Record Dates: First submitted 2013-04-02; First posted 2013-05-17 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Prophylaxis of A/H3N2v Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): 3.75 µg H3N2c HA + 0.125 mL MF59
  Interventions: Biological: Swine Influenza
- Group B (Experimental): 7.5 µg H3N2c HÁ + 0.250 mL MF59
  Interventions: Biological: Swine Influenza
- Group C (Experimental): 15 µg H3N2c unadjuvanted
  Interventions: Biological: Swine Influenza

INTERVENTIONS:
Biological: Swine Influenza — Comparison of different dosages of vaccines

SUMMARY:
Evaluate the safety and immunogenicity of three dosage levels of swine influenza vaccine in children ages 3 to <9 years, adolescents 9 to <18 years, adults 18 to <65 years and elderly 65 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 3 years of age and older
2. Individuals or, (for children and adolescents) parents or legal guardians, who have given written consent after the nature of the study has been explained according to local regulatory requirements. Assent is required depending on age of child/adolescent
3. Individuals in good health as determined by the outcome of medical history, physical examination, and clinical judgment of the investigator
4. Individuals who can comply with study procedures and are available for follow-up

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment, including psychiatric illness, as determined by the investigator's clinical judgement may interfere with the subject's ability to participate in study
2. Individuals with any progressive or severe neurologic disorder, seizure disorder or recent history of Guillian-Barré syndrome
3. Individuals or (for children and adolescents) parents or legal guardians who are not able to comprehend and to follow all required study procedures for the whole period of the study
4. Individuals with a history of illness/with an ongoing illness that, in the opinion of the investigator, may pose additional risk to the subject if he/she participates in the study
5. Individuals who have a suspected/confirmed diagnosis for any Adverse event of Special interest
6. Individuals with known or suspected impairment of the immune system including, but not limited to:

   * autoimmune disease such as rheumatoid arthritis, HIV infection, hypo- or agammaglobulinemia;
   * autoimmune disorders;
   * Systemic therapy with corticosteroids or other immunosuppressive therapy.
   * Receipt of immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Day 1 or planned during the full length of the study
7. Individuals who are pregnant or breastfeeding. Female subjects of childbearing potential must have a negative pregnancy test prior to study vaccines being administered
8. If female, "of childbearing potential", sexually active, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to study entry
9. "Of childbearing potential" is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy
10. Acceptable birth control methods are defined as one or more of the following:

    1. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring);
    2. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse;
    3. Intrauterine device (IUD);
    4. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the subject's study entry.
11. If female of childbearing potential and sexually active, refusal to use an "acceptable contraceptive method" through to 3 weeks after last study vaccination
12. Individuals who are allergic to any of the vaccine components.
13. For children 17 years of age and younger: Individuals who have had ever a malignancy
14. For adults 18 years or older: Individuals who have had a malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder within the past 5 years
15. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study
16. Individuals with a body temperature >38°C (>100.4°F) or any acute illness within 3 days of intended study vaccination
17. Individuals who have had a previous confirmed or suspected illness from swine flu (H3N2v)
18. Individuals who have received any prior H3N2v vaccine
19. Individuals who have received any other type of influenza vaccination (e.g., "seasonal") within 14 days prior to enrolment, or who plans to receive influenza vaccine during the treatment phase of this study (seasonal influenza vaccination is allowed after Day 43/Visit 3)
20. Individuals who received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study or who are planning to receive any (non-influenza) vaccine within 4 weeks from the study vaccines
21. Individuals who are research staff involved with the clinical study or family/household members of research staff
22. Individuals with a BMI > 35 kg/m2 (adults), > 29 kg/m2 (adolescents), or > 21 kg/m2 (children)
23. Individuals with a history of drug or alcohol abuse within the past 2 years

Ages: 3 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (11):
- United States (11):
  - 51, Northern California Clinical Research Center, Redding, California
  - 47, Benchmark Research, Sacramento, California
  - 46, Johnson County Clinical Trials, Lenexa, Kansas
  - 49, Heartland Research Associates, LLC, Wichita, Kansas
  - 43, Central Kentucky Research Associates, Lexington, Kentucky
  - 41, Benchmark Research, Metairie, Louisiana
  - 44, Rochester Clinical Research Inc., Rochester, New York
  - 50, PMG Research of Raleigh, Raleight, North Carolina
  - 45, Omega Medical Research, Warwick, Rhode Island
  - 42, Research Acros, Dallas, Texas
  - 48, "J. Lewis Research, Inc., Salt Lake City, Utah

REFERENCES:
- [Derived] Johnson C, Hohenboken M, Poling T, Jaehnig P, Kanesa-Thasan N. Safety and Immunogenicity of Cell Culture-Derived A/H3N2 Variant Influenza Vaccines: A Phase I Randomized, Observer-Blind, Dose-Ranging Study. J Infect Dis. 2015 Jul 1;212(1):72-80. doi: 10.1093/infdis/jiu826. Epub 2014 Dec 23. PMID 25538277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 11 study centres in USA.
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 Age Group: 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C Age Group: 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 Age Group: ≥65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 Age Group: ≥65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C Age Group: ≥65 YEARS: Subjects ≥65 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Period: Overall Study
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥65 YEARS | A/H3N2C + MF59 Age Group: ≥65 YEARS | A/H3N2C Age Group: ≥65 YEARS
Started | 54 | 55 | 51 | 53 | 51 | 53 | 53 | 55 | 48 | 51 | 51 | 52
Completed | 38 | 44 | 39 | 49 | 50 | 50 | 43 | 47 | 46 | 49 | 46 | 49
Not Completed | 16 | 11 | 12 | 4 | 1 | 3 | 10 | 8 | 2 | 2 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 10 | 7 | 3 | 0 | 3 | 4 | 7 | 2 | 0 | 0 | 2
Not completed — Other - Unclassified | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 4 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis was done on all enrolled set.
Groups:
- A/H3N2C + 1/2 MF59 : 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 : 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C : 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 : 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 : 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C : 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 : 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 : 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C : 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 : ≥65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 : ≥65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C : ≥65 YEARS: Subjects ≥65 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- Total: Total of all reporting groups
Arm/Group | A/H3N2C + 1/2 MF59 : 3 TO <9 YEARS | A/H3N2C + MF59 : 3 TO <9 YEARS | A/H3N2C : 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 : 9 TO <18 YEARS | A/H3N2C + MF59 : 9 TO <18 YEARS | A/H3N2C : 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 : 18 TO <65 YEARS | A/H3N2C + MF59 : 18 TO <65 YEARS | A/H3N2C : 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 : ≥65 YEARS | A/H3N2C + MF59 : ≥65 YEARS | A/H3N2C : ≥65 YEARS | Total
Number analyzed (Participants) | 54 | 55 | 51 | 53 | 51 | 53 | 53 | 55 | 48 | 51 | 51 | 52 | 627
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 6 (1.7) | 6 (1.6) | 6.2 (1.6) | 12.6 (2.7) | 12.8 (2.4) | 12.3 (2.4) | 42.3 (12.8) | 42.4 (13.3) | 44 (14.9) | 71.3 (5.3) | 72.9 (6.1) | 73.8 (6.1) | 33.2 (27.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 26 | 29 | 25 | 26 | 32 | 25 | 28 | 31 | 25 | 32 | 336
  Male | 24 | 28 | 25 | 24 | 26 | 27 | 21 | 30 | 20 | 20 | 26 | 20 | 291

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects (3 to <9 Years of Age) Reporting Solicited Adverse Events (AEs) Following Vaccination With H3N2 Monovalent Vaccine.
Description: Safety and tolerability of H3N2 monovalent vaccine was assessed in terms of the number of subjects (3 to <9 years of age) reporting solicited local and systemic adverse events and other adverse events after each vaccination.
Time Frame: Day 1 through Day 7 after each vaccination
Population: Analysis was done on Solicited Safety Set.
Measure: Number; unit: Number of Subjects
Groups:
- A/H3N2C + 1/2 MF59 - Age Group: 3 TO <9 YEARS: Subjects, 3 to < 9 years old, received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 - Age Group: 3 TO <9 YEARS: Subjects, 3 to < 9 years old, received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg antigen adjuvanted with full dose MF59.
- A/H3N2C - Age Group: 3 TO <9 YEARS: Subjects, 3 to < 9 years old, received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Arm/Group | A/H3N2C + 1/2 MF59 - Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 - Age Group: 3 TO <9 YEARS | A/H3N2C - Age Group: 3 TO <9 YEARS
Number analyzed (Participants) | 49 | 53 | 49
Number of Subjects
  ANY- Vac. 1 | 31 | 36 | 18
  ANY- Vac. 2 (N= 45,52,48) | 24 | 25 | 22
  INJECTION SITE REACTIONS- Vacc. 1 | 28 | 33 | 16
  INJECTION SITE REACTIONS- Vacc. 2 | 22 | 24 | 17
  ECCHYMOSIS (mm), < 6y (T.II, 1st Vac.,N=14,20,15) | 2 | 0 | 0
  ECCHYMOSIS (mm), < 6y (T.II, 2nd Vac.,N=11,21,16) | 1 | 2 | 0
  ECCHYMOSIS (mm), ≥ 6y (T.II, 1st Vac.,N=33,29,31) | 0 | 0 | 0
  ECCHYMOSIS (mm), ≥ 6y (T.II, 2nd Vac.,N=32,31,32) | 0 | 0 | 0
  ERYTHEMA (mm), < 6y (T.II, 1st Vac.,N=14,20,16) | 1 | 1 | 0
  ERYTHEMA (mm), ≥ 6y (T.II, 1st Vac.,N=33,29,31) | 2 | 0 | 1
  ERYTHEMA (mm), < 6y (T.II, 2nd Vac.,N=12,21,16) | 0 | 2 | 0
  ERYTHEMA (mm), ≥ 6y (T.II, 2nd Vac.,N=31,31,31) | 2 | 1 | 0
  INDURATION (mm), < 6y (T.II, 1st Vac.,N=14,20,16) | 0 | 1 | 0
  INDURATION (mm), < 6y (T.II, 2nd Vac.,N=12,21,16) | 0 | 1 | 0
  INDURATION (mm), ≥ 6y (T.II, 1st Vac.,N=33,29,32) | 2 | 3 | 0
  INDURATION (mm), ≥ 6y (T.II, 2nd Vac.,N=32,31,31) | 1 | 1 | 0
  SYSTEMIC REACTIONS- Vacc. 1 | 15 | 19 | 7
  SYSTEMIC REACTIONS- Vacc. 2 | 16 | 11 | 12
  ARTHRALGIA (1st Vac.,N=31,27,30) | 1 | 1 | 1
  ARTHRALGIA (2nd Vac.,N=33,29,31) | 1 | 0 | 0
  BODY TEMPERATURE ≥38°C (1st Vac.,N=49,53,49) | 0 | 1 | 0
  BODY TEMPERATURE ≥38°C (2nd Vac.,N=42,52,48) | 0 | 2 | 0
  CHANGE IN EATING HABITS (1st Vac.,N=13,19,15) | 1 | 1 | 0
  CHANGE IN EATING HABITS (2nd Vac.,N=12,20,16) | 1 | 3 | 1
  DIARRHEA (1st Vac.,N=45,46,46) | 0 | 3 | 0
  DIARRHEA (2nd Vac.,N=43,50,46) | 1 | 1 | 1
  FATIGUE (1st Vac.,N=31,28,31) | 5 | 9 | 4
  FATIGUE (2nd Vac.,N=33,30,32) | 5 | 1 | 3
  HEADACHE (1st Vac.,N=32,28,31) | 6 | 5 | 3
  HEADACHE (2nd Vac.,N=33,31,32) | 4 | 4 | 2
  IRRITABILITY (1st Vac.,N=13,19,16) | 2 | 2 | 1
  IRRITABILITY (2nd Vac.,N=11,20,16) | 3 | 3 | 3
  LOSS OF APPETITE (1st Vac.,N=32,27,32) | 2 | 2 | 1
  LOSS OF APPETITE (2nd Vac.,N=32,30,30) | 4 | 1 | 2
  MALAISE (1st Vac.,N=32,28,32) | 4 | 7 | 0
  MALAISE (2nd Vac.,N=32,30,30) | 6 | 4 | 3
  MYALGIA (1st Vac.,N=32,28,32) | 3 | 2 | 1
  MYALGIA (2nd Vac.,N=33,31,32) | 4 | 1 | 1
  NAUSEA (1st Vac.,N=32,28,31) | 5 | 2 | 1
  NAUSEA (2nd Vac.,N=31,31,30) | 3 | 2 | 1
  PREV.OF PAIN/FEVER (1st Vac.,N=46,48,46) | 0 | 1 | 1
  PREV.OF PAIN/FEVER (2nd Vac.,N=44,51,47) | 1 | 0 | 2
  SLEEPINESS (1st Vac.,N=13,19,16) | 2 | 2 | 1
  SLEEPINESS (2nd Vac.,N=12,20,16) | 1 | 3 | 1
  TREAT.OF PAIN/FEVER (1st Vac.,N=46,49,46) | 4 | 6 | 2
  TREAT.OF PAIN/FEVER (2nd Vac.,N=44,51,47) | 1 | 2 | 3
  VOMITING (1st Vac.,N=46,47,48) | 1 | 3 | 0
  VOMITING (2nd Vac.,N=44,51,46) | 2 | 2 | 3

2. Primary Outcome: Number of Subjects (9 to <18 Years of Age) Reporting Solicited Adverse Events Following Vaccination With H3N2 Monovalent Vaccine.
Description: Safety and tolerability of H3N2 monovalent vaccine was assessed in terms of the number of subjects (9 to <18 years of age) reporting solicited local and systemic adverse events and other adverse events after each vaccination.
Time Frame: Day 1 through Day 7 after each vaccination
Population: Analysis was done on Solicited Safety Set.
Measure: Number; unit: Number of Subjects
Groups:
- A/H3N2C + 1/2 MF59 - Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75µg antigen adjuvanted with half dose MF59 Subjects 3 to <9 years.
- A/H3N2C + MF59 - Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C - Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Arm/Group | A/H3N2C + 1/2 MF59 - Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 - Age Group: 9 TO <18 YEARS | A/H3N2C - Age Group: 9 TO <18 YEARS
Number analyzed (Participants) | 54 | 51 | 53
Number of Subjects
  ANY- Vac. 1 | 37 | 40 | 35
  ANY- Vac. 2 (N=52,48,53) | 30 | 24 | 27
  INJECTION SITE REACTIONS- Vacc. 1 | 35 | 34 | 27
  INJECTION SITE REACTIONS- Vacc. 2 | 24 | 20 | 23
  ECCHYMOSIS (mm), ≥ 6y (T.II, 1st Vac.,N=53,51,53) | 0 | 1 | 0
  ECCHYMOSIS (mm), ≥ 6y (T.II) (2nd Vac.,N=52,48,52) | 0 | 1 | 0
  ERYTHEMA (mm), ≥ 6y (T.II) (1st Vac.,N=52,51,53) | 0 | 3 | 1
  ERYTHEMA (mm), ≥ 6y (T.II) (2nd Vac.,N=51,48,52) | 1 | 2 | 1
  INDURATION (mm), ≥ 6y (T.II) (1st Vac.,N=52,51,53) | 2 | 7 | 2
  INDURATION (mm), ≥ 6y (T.II) (2nd Vac.,N=52,48,52) | 3 | 4 | 1
  SYSTEMIC REACTIONS- Vacc. 1 | 25 | 32 | 26
  SYSTEMIC REACTIONS- Vacc. 2 | 17 | 14 | 15
  ARTHRALGIA (1st Vac.,N=51,50,51) | 3 | 3 | 7
  ARTHRALGIA (2nd Vac.,N=49,48,52) | 4 | 1 | 2
  BODY TEMPERATURE >=38C (1st Vac.,N=53,51,53) | 0 | 1 | 1
  BODY TEMPERATURE ≥38°C (2nd Vac.,N=51,48,52) | 0 | 1 | 0
  DIARRHEA (1st Vac.,N=51,51,51) | 3 | 5 | 2
  DIARRHEA (2nd Vac.,N=50,47,49) | 2 | 2 | 4
  FATIGUE (1st Vac.,N=53,51,53) | 12 | 16 | 18
  FATIGUE (2nd Vac.,N=51,48,53) | 9 | 12 | 9
  HEADACHE (1st Vac.,N=53,50,53) | 13 | 16 | 11
  HEADACHE (2nd Vac.,N=50,48,53) | 11 | 9 | 9
  LOSS OF APPETITE (1st Vac.,N=53,51,51) | 6 | 9 | 6
  LOSS OF APPETITE (2nd Vac.,N=51,48,49) | 5 | 4 | 2
  MALAISE (1st Vac.,N=53,51,51) | 10 | 12 | 10
  MALAISE (2nd Vac.,N=51,48,49) | 7 | 5 | 4
  MYALGIA (1st Vac.,N=52,51,53) | 6 | 9 | 5
  MYALGIA (2nd Vac.,N=50,48,53) | 5 | 2 | 2
  NAUSEA (1st Vac.,N=53,51,53) | 9 | 10 | 5
  NAUSEA (2nd Vac.,N=50,48,53) | 3 | 3 | 6
  PREV.OF PAIN/FEVER (1st Vac.,N=54,49,52) | 0 | 3 | 0
  PREV.OF PAIN/FEVER (2nd Vac.,N=50,47,53) | 0 | 1 | 1
  TREAT.OF PAIN/FEVER (1st Vac.,N=54,50,52) | 5 | 4 | 2
  TREAT.OF PAIN/FEVER (2nd Vac.,N=49,47,53) | 3 | 2 | 1
  VOMITING (1st Vac.,N=53,51,51) | 2 | 1 | 0
  VOMITING (2nd Vac.,N=50,48,49) | 1 | 0 | 0

3. Primary Outcome: Number of Subjects (18 to < 65 Years) Reporting Solicited Adverse Events Following Vaccination With H3N2 Monovalent Vaccine.
Description: Safety and tolerability of H3N2 monovalent vaccine was assessed in terms of the number of subjects (18 to < 65 years of age) reporting solicited local and systemic adverse events and other adverse events after each vaccination.
Time Frame: Day 1 through Day 7 after each vaccination
Population: Analysis was done on Solicited Safety Set.
Measure: Number; unit: Number of Subjects
Groups:
- A/H3N2C + 1/2 MF59 - Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 - Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C - Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old Received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Arm/Group | A/H3N2C + 1/2 MF59 - Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 - Age Group: 18 TO <65 YEARS | A/H3N2C - Age Group: 18 TO <65 YEARS
Number analyzed (Participants) | 51 | 54 | 48
Number of Subjects
  ANY- Vac. 1 | 30 | 40 | 27
  ANY- Vac. 2 (N=47,51,48) | 21 | 28 | 21
  INJECTION SITE REACTIONS- Vacc. 1 | 23 | 32 | 19
  INJECTION SITE REACTIONS- Vacc. 2 | 17 | 24 | 15
  ECCHYMOSIS (mm), ≥ 6y (T.II, 1st Vac.,N=50,52,45) | 0 | 1 | 0
  ECCHYMOSIS (mm), ≥ 6y (T.II, 2nd Vac.,N=46,51,48) | 0 | 0 | 1
  ERYTHEMA (mm), ≥ 6y (T.II, 1st Vac.,N=50,53,47) | 0 | 5 | 0
  ERYTHEMA (mm), ≥ 6y (T.II, 2nd Vac.,N=46,50,48) | 0 | 1 | 0
  INDURATION (mm), ≥ 6y (T.II, 1st Vac.,N=50,53,46) | 1 | 8 | 1
  INDURATION (mm), ≥ 6y (T.II, 2nd Vac.,N=46,51,48) | 1 | 2 | 0
  SYSTEMIC REACTIONS- Vacc. 1 | 23 | 27 | 19
  SYSTEMIC REACTIONS- Vacc. 2 | 15 | 20 | 13
  ARTHRALGIA (1st Vac.,N=50,51,45) | 4 | 5 | 3
  ARTHRALGIA (2nd Vac.,N=46,48,48) | 3 | 4 | 5
  BODY TEMPERATURE ≥38°C (1st Vac.,N=51,54,47) | 2 | 1 | 0
  BODY TEMPERATURE ≥38°C (2nd Vac.,N=47,50,47) | 0 | 0 | 0
  DIARRHEA (1st Vac.,N=49,52,46) | 6 | 10 | 3
  DIARRHEA (2nd Vac.,N=44,50,47) | 4 | 6 | 1
  FATIGUE (1st Vac.,N=50,53,47) | 10 | 11 | 8
  FATIGUE (2nd Vac.,N=45,48,48) | 7 | 8 | 7
  HEADACHE (1st Vac.,N=51,53,47) | 11 | 11 | 10
  HEADACHE (2nd Vac.,N=47,49,48) | 9 | 9 | 8
  LOSS OF APPETITE (1st Vac.,N=50,53,47) | 4 | 4 | 4
  LOSS OF APPETITE (2nd Vac.,N=46,50,47) | 0 | 4 | 1
  MALAISE (1st Vac.,N=49,53,47) | 12 | 12 | 4
  MALAISE (2nd Vac.,N=45,50,47) | 3 | 10 | 4
  MYALGIA (1st Vac.,N=51,51,45) | 7 | 7 | 6
  MYALGIA (2nd Vac.,N=47,48,48) | 2 | 5 | 4
  NAUSEA (1st Vac.,N=50,52,47) | 3 | 5 | 3
  NAUSEA (2nd Vac.,N=47,50,47) | 3 | 5 | 2
  PREV.OF PAIN/FEVER (1st Vac.,N=49,52,48) | 0 | 0 | 0
  PREV.OF PAIN/FEVER (2nd Vac.,N=46,50,46) | 0 | 1 | 0
  TREAT.OF PAIN/FEVER (1st Vac.,N=49,53,48) | 5 | 4 | 1
  TREAT.OF PAIN /FEVER (2nd Vac.,N=46,50,46) | 1 | 2 | 0
  VOMITING (1st Vac.,N=49,53,47) | 0 | 0 | 2
  VOMITING (2nd Vac.,N=46,50,47) | 0 | 1 | 1

4. Primary Outcome: Number of Subjects (≥ 65 Years) Reporting Solicited Adverse Events Following Vaccination With H3N2 Monovalent Vaccine.
Description: Safety and tolerability of H3N2 monovalent vaccine was assessed in terms of the number of subjects (≥ 65 years of age) reporting solicited local and systemic adverse events and other adverse events after each vaccination.
Time Frame: Day 1 through Day 7 after each vaccination
Population: Analysis was done on Solicited Safety Set.
Measure: Number; unit: Number of Subjects
Groups:
- A/H3N2C + 1/2 MF59 - Age Group: ≥65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 - Age Group: ≥65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg antigen adjuvanted with full dose MF59.
- A/H3N2C - Age Group: ≥65 YEARS: Subjects ≥65 years old Received two injections of cell-culture derived H3N2c vaccine, each dose containing 15 µg H3N2c antigen.
Arm/Group | A/H3N2C + 1/2 MF59 - Age Group: ≥65 YEARS | A/H3N2C + MF59 - Age Group: ≥65 YEARS | A/H3N2C - Age Group: ≥65 YEARS
Number analyzed (Participants) | 51 | 49 | 50
Number of Subjects
  ANY- Vac. 1 | 23 | 29 | 15
  ANY- Vac. 2 (N=51,45,48) | 14 | 17 | 14
  INJECTION SITE REACTIONS- Vac. 1 | 11 | 21 | 6
  INJECTION SITE REACTIONS- Vac. 2 | 9 | 14 | 5
  ECCHYMOSIS (mm), ≥ 6y (T.II, 1st Vac.,N=51,49,50) | 2 | 0 | 0
  ECCHYMOSIS (mm), ≥ 6y (T.II, 2nd Vac.,N=49,45,48) | 0 | 0 | 1
  ERYTHEMA (mm), ≥ 6y (T.II, 1st Vac.,N=51,45,49) | 1 | 1 | 2
  ERYTHEMA (mm), ≥ 6y (T.II, 2nd Vac.,N=49,44,48) | 1 | 2 | 1
  INDURATION (mm), ≥ 6y (T.II, 1st Vac.,N=51,48,50) | 1 | 2 | 2
  INDURATION (mm), ≥ 6y (T.II, 2nd Vac.,N=49,44,48) | 0 | 2 | 1
  SYSTEMIC REACTIONS- Vacc. 1 | 17 | 16 | 13
  SYSTEMIC REACTIONS- Vacc. 2 | 8 | 11 | 11
  ARTHRALGIA (1st Vac.,N=47,45,50) | 3 | 4 | 3
  ARTHRALGIA (2nd Vac.,N=50,43,47) | 3 | 1 | 2
  BODY TEMPERATURE ≥38°C (1st Vac.,N=51,48,50) | 0 | 0 | 0
  BODY TEMPERATURE ≥38°C (2nd Vac.,N=51,44,48) | 0 | 0 | 1
  DIARRHEA (1st Vac.,N=50,47,48) | 5 | 3 | 4
  DIARRHEA (2nd Vac.,N=49,44,44) | 2 | 1 | 1
  FATIGUE (1st Vac.,N=49,48,49) | 8 | 8 | 4
  FATIGUE (2nd Vac.,N=51,44,48) | 5 | 6 | 3
  HEADACHE (1st Vac.,N=50,49,50) | 8 | 6 | 4
  HEADACHE (2nd Vac.,N=51,44,48) | 5 | 2 | 3
  LOSS OF APPETITE (1st Vac.,N=50,48,49) | 6 | 2 | 2
  LOSS OF APPETITE (2nd Vac.,N=50,45,46) | 3 | 1 | 1
  MALAISE (1st Vac.,N=50,48,49) | 5 | 6 | 2
  MALAISE (2nd Vac.,N=50,45,46) | 4 | 3 | 1
  MYALGIA (1st Vac.,N=49,48,50) | 4 | 5 | 3
  MYALGIA (2nd Vac.,N=50,43,48) | 2 | 1 | 3
  NAUSEA (1st Vac.,N=51,49,50) | 5 | 3 | 3
  NAUSEA (2nd Vac.,N=50,45,47) | 2 | 2 | 1
  PREV.OF PAIN/FEVER (1st Vac.,N=48,46,50) | 1 | 0 | 0
  PREV.OF PAIN/FEVER (2nd Vac.,N=50,44,48) | 0 | 0 | 0
  TREAT.OF PAIN/FEVER (1st Vac.,N=48,46,50) | 0 | 3 | 1
  TREAT.OF PAIN/FEVER (2nd Vac.,N=50,44,48) | 0 | 1 | 3
  VOMITING (1st Vac.,N=51,48,49) | 0 | 0 | 1
  VOMITING (2nd Vac.,N=49,45,46) | 0 | 0 | 0

5. Primary Outcome: Number of Subjects (3 to ≥ 65 Years of Age) Reporting Unsolicited Adverse Events Following Vaccination With H3N2 Monovalent Vaccine.
Description: The number of subjects reporting any unsolicited adverse events (AEs) from day 1 through day 21 after last vaccination within each vaccine group are reported.
  The number of subjects reporting any serious adverse events (SAEs), AEs leading to withdrawal from the study, medically attended AEs, AE of special interest (AESI), new onset chronic disease (NOCDs) from day 1 through day 366, after receiving with H3N2 monovalent vaccine are reported.
Time Frame: Day 1 through Day 366
Population: Analysis was done on unsolicited safety dataset i.e. all subjects in the exposed population who have post-vaccination unsolicited adverse event records.
Measure: Number; unit: Number of subjects
Groups:
- A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75µg antigen adjuvanted with half dose MF59.
- A/H3N2C Age Group: 3 TO <9 YEARS: Subjects 3 to <9 years old received two injections of of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 Age Group: >=65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 Age Group: >=65 YEARS: Subjects ≥65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C Age Group: >=65 YEARS: Subjects ≥65 years old received two injections of of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: >=65 YEARS | A/H3N2C + MF59 Age Group: >=65 YEARS | A/H3N2C Age Group: >=65 YEARS
Number analyzed (Participants) | 50 | 54 | 50 | 54 | 51 | 53 | 51 | 54 | 48 | 52 | 49 | 51
Number of subjects
  Any AE (Day 1 to Day 366) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 5 | 5
  At least possibly related AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 5 | 5
  At least possibly related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE leading to withdrawal | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 3 | 1
  Medically attended AEs | 8 | 21 | 14 | 13 | 13 | 20 | 21 | 17 | 13 | 31 | 22 | 23
  AESI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NOCD | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 3 | 1 | 7 | 1 | 6
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Percentages of Subjects (3 to ≥ 65 Years of Age) With Seroconversion or Significant Increase in Hemagglutination Inhibition (HI) Antibody Titers Following Vaccination With H3N2 Monovalent Vaccine.
Description: The percentages of subjects (3 to ≥ 65 years of age) achieving seroconversion or significant increase in HI antibody titers against H3N2 homologous strain, three weeks after receiving first (Day 22) and second (Day 43) vaccination are reported.
  Seroconversion is defined as HI titer ≥1:40 for subjects negative at baseline (HI titer <1:10); or a minimum 4-fold increase in HI titer for subjects positive at baseline (HI titer ≥1:10) on Day 22 and Day 43.
Time Frame: Day 22, Day 43 post vaccination
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS: Subjects 9 to <18 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS: Subjects 18 to <65 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥65 YEARS | A/H3N2C + MF59 Age Group: ≥65 YEARS | A/H3N2C Age Group: ≥65 YEARS
Number analyzed (Participants) | 47 | 54 | 49 | 52 | 49 | 53 | 52 | 54 | 48 | 49 | 49 | 51
Percentages of Subjects
  Day 22 (N=47,54,49,52,48,53,52,54,48,49,49,51) | 96 [85.5 to 99.5] | 98 [90.1 to 99.95] | 71 [56.7 to 83.4] | 88 [76.6 to 95.6] | 98 [88.9 to 99.95] | 85 [72.4 to 93.3] | 73 [59 to 84.4] | 89 [77.4 to 95.8] | 67 [51.6 to 79.6] | 57 [42.2 to 71.2] | 71 [56.7 to 83.4] | 61 [46.1 to 74.2]
  Day 43(N=43,53,48,52,49,53,51,52,48,48,49,50) | 100 [91.8 to 100] | 100 [93.3 to 100] | 92 [80 to 97.7] | 94 [84.1 to 98.8] | 98 [89.1 to 99.95] | 91 [79.3 to 96.9] | 82 [69.1 to 91.6] | 92 [81.5 to 97.9] | 71 [55.9 to 83] | 58 [43.2 to 72.4] | 80 [65.7 to 89.8] | 64 [49.2 to 77.1]

7. Secondary Outcome: Geometric Mean HI Antibody Titers (GMTs) Following Vaccination With H3N2 Monovalent Vaccine (3 to ≥ 65 Years of Age).
Description: The HI antibody titers against H3N2 homologous strain at baseline (Day 1), three weeks after first (Day 22) and second (Day 43) vaccination and persisting titers at six months (Day 183) and one year (Day 366) after vaccination are reported in terms of GMTs is reported across subjects with age groups 3 to ≥ 65 years.
Time Frame: Day 1, Day 22, Day 43, Day 183 and Day 366 post vaccination
Population: Analysis was done on Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥65 YEARS | A/H3N2C + MF59 Age Group: ≥65 YEARS | A/H3N2C Age Group: ≥65 YEARS
Number analyzed (Participants) | 53 | 55 | 50 | 53 | 51 | 53 | 53 | 55 | 48 | 50 | 50 | 52
Titers
  Day 1 | 8.48 [6.89 to 10] | 8.26 [6.74 to 10] | 8.8 [7.10 to 11] | 28 [21 to 37] | 29 [22 to 39] | 27 [20 to 35] | 34 [26 to 44] | 52 [40 to 68] | 42 [32 to 56] | 36 [28 to 47] | 32 [25 to 42] | 26 [20 to 34]
  Day 22 (N=47,54,49,52,48,53,52,54,48,49,49,51) | 192 [134 to 275] | 277 [198 to 387] | 93 [65 to 132] | 386 [293 to 510] | 456 [341 to 609] | 343 [261 to 452] | 300 [217 to 415] | 504 [367 to 692] | 226 [162 to 315] | 135 [103 to 177] | 206 [157 to 270] | 140 [107 to 183]
  Day 43 (N=43,53,48,52,49,53,51,52,48,48,49,50) | 524 [396 to 694] | 679 [527 to 874] | 198 [152 to 258] | 486 [379 to 623] | 656 [508 to 849] | 389 [304 to 498] | 276 [208 to 365] | 427 [324 to 564] | 261 [196 to 347] | 131 [102 to 170] | 202 [157 to 261] | 163 [126 to 210]
  Day 183 (N=39,44,42,47,50,47,45,50,46,47,48,49) | 97 [75 to 126] | 145 [113 to 185] | 67 [52 to 86] | 173 [137 to 218] | 242 [194 to 302] | 170 [135 to 214] | 161 [120 to 217] | 219 [166 to 289] | 188 [142 to 251] | 93 [72 to 121] | 122 [94 to 157] | 98 [76 to 126]
  Day 366 (N=38,43,38,47,50,47,43,47,46,48,46,49) | 46 [35 to 61] | 70 [53 to 91] | 37 [28 to 49] | 112 [86 to 148] | 124 [96 to 161] | 111 [84 to 145] | 111 [84 to 148] | 170 [130 to 223] | 126 [96 to 165] | 55 [43 to 69] | 71 [56 to 91] | 68 [53 to 86]

8. Secondary Outcome: Geometric Mean Ratio of Subjects (3 to ≥ 65 Years of Age) Post Versus Pre-vaccination HI Antibody Titers Following Vaccination With H3N2 Monovalent Vaccine.
Description: The geometric mean ratio (GMR) of post versus pre-vaccination HI antibody titers against H3N2 homologous strain following vaccination as compared to baseline titers are reported for after first (Day 22/Day 1) and second (Day 43/Day 1) vaccination and for persisting titers at six months (Day 183/Day1) and one year (Day 366/Day 1) is reported across subjects with age groups 3 to ≥ 65 years.
Time Frame: Day 22/Day 1, Day 43/Day 1, Day 183/Day 1, Day 366/Day 1
Population: Analysis was done on Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥65 YEARS | A/H3N2C + MF59 Age Group: ≥65 YEARS | A/H3N2C Age Group: ≥65 YEARS
Number analyzed (Participants) | 47 | 54 | 49 | 52 | 48 | 53 | 52 | 54 | 48 | 49 | 49 | 51
Ratios
  Day22/Day1 | 22 [15 to 32] | 33 [23 to 47] | 11 [7.51 to 16] | 14 [9.58 to 19] | 15 [10 to 22] | 13 [8.91 to 18] | 7.54 [5.41 to 11] | 11 [8.16 to 16] | 5.35 [3.80 to 7.55] | 3.79 [2.71 to 5.29] | 6.64 [4.75 to 9.28] | 5.13 [3.70 to 7.13]
  Day43/Day1 (N=43,53,48,52,49,53,51,52,48,48,49,50) | 59 [43 to 81] | 82 [62 to 109] | 23 [17 to 31] | 18 [13 to 25] | 21 [15 to 30] | 14 [10 to 20] | 7.16 [5.34 to 9.61] | 9.58 [7.17 to 13] | 6.24 [4.62 to 8.44] | 3.82 [2.80 to 5.21] | 6.55 [4.81 to 8.91] | 5.94 [4.38 to 8.07]
  Day183/Day1(N=39,44,42,47,50,47,45,50,46,47,48,49) | 10 [7.48 to 14] | 17 [13 to 23] | 7.17 [5.31 to 9.68] | 6.59 [4.87 to 8.91] | 8.2 [6.13 to 11] | 6.38 [4.73 to 8.63] | 3.95 [2.93 to 5.31] | 4.95 [3.75 to 6.54] | 4.4 [3.29 to 5.87] | 2.6 [1.93 to 3.49] | 3.83 [2.85 to 5.14] | 3.4 [2.54 to 4.55]
  Day366/Day1(N=38,43,38,47,50,47,43,47,46,48,46,49) | 4.83 [3.43 to 6.79] | 8.23 [5.98 to 11] | 4.13 [2.93 to 5.82] | 4.28 [3.07 to 5.95] | 4.21 [3.06 to 5.79] | 4.15 [2.99 to 5.77] | 2.79 [2.10 to 3.70] | 3.97 [3.03 to 5.21] | 2.99 [2.28 to 3.93] | 1.6 [1.23 to 2.09] | 2.33 [1.77 to 3.05] | 2.33 [1.79 to 3.03]

9. Secondary Outcome: Percentages of Subjects (3 to ≥ 65 Years of Age) Achieving HI Titers ≥1:40 Following Vaccination With H3N2 Monovalent Vaccine.
Description: The percentages of subjects (3 to ≥ 65 years of age) demonstrating HI titers ≥1:40 against H3N2 homologous strain on Day 183 and Day 366 post vaccination.
Time Frame: Day 183 and Day 366 post vaccination
Population: Analysis was done on the full analysis set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- A/H3N2C Age Group: ≥65 YEARS: Subjects ≥65 years old received two injections of of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥65 YEARS | A/H3N2C + MF59 Age Group: ≥65 YEARS | A/H3N2C Age Group: ≥65 YEARS
Number analyzed (Participants) | 39 | 44 | 42 | 47 | 50 | 47 | 45 | 50 | 46 | 48 | 48 | 49
Percentages of Subjects
  Day 183 (N=39,44,42,47,50,47,45,50,46,47,48,49) | 95 [82.7 to 99.4] | 98 [88 to 99.94] | 81 [65.9 to 91.4] | 98 [88.7 to 99.95] | 100 [92.9 to 100] | 100 [92.5 to 100] | 87 [73.2 to 94.9] | 100 [92.9 to 100] | 87 [73.7 to 95.1] | 91 [79.6 to 97.6] | 94 [82.8 to 98.7] | 88 [75.2 to 95.4]
  Day 366 (N=38,43,38,47,50,47,43,47,46,48,46,49) | 82 [65.7 to 92.3] | 91 [77.9 to 97.4] | 58 [40.8 to 73.7] | 94 [82.5 to 98.7] | 98 [89.4 to 99.95] | 89 [76.9 to 96.5] | 81 [66.6 to 91.6] | 96 [85.5 to 99.5] | 80 [66.1 to 90.6] | 75 [60.4 to 86.4] | 80 [66.1 to 90.6] | 80 [65.7 to 89.8]

10. Secondary Outcome: Percentages of Subjects (3 to ≥ 61 Years of Age) With Seroconversion or Significant Increase in Hemagglutination Inhibition Antibody Titers Following Vaccination With H3N2 Monovalent Vaccine.
Description: The percentage of subjects achieving seroconversion or significant increase for HI antibody titers at three weeks after receiving first (Day 22) and second (Day 43) vaccination is reported, across age groups of 3 to ≥61 years.
  Seroconversion is defined as HI titer ≥1:40 for subjects negative at baseline (HI titer <1:10); or a minimum 4-fold increase in HI titer for subjects positive at baseline (HI titer ≥1:10) on Day 22 and Day 43.
Time Frame: Day 22, Day 43 post vaccination
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- A/H3N2C + 1/2 MF59 Age Group: 18 TO <61 YEARS: Subjects 18 to <61 years old Received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 Age Group: 18 TO <61 YEARS: Subjects 18 to <61 years old Received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C Age Group: 18 TO <61 YEARS: Subjects 18 to <61 years old Received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 Age Group: ≥61 YEARS: Subjects ≥61 years old Received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C + MF59 Age Group: ≥61 YEARS: Subjects ≥61 years old Received two injections of cell-culture derived H3N2c vaccine, each dose containing 7.5 µg H3N2c antigen adjuvanted with full dose MF59.
- A/H3N2C Age Group: ≥61 YEARS: Subjects ≥61 years old Received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <61 YEARS | A/H3N2C + MF59 Age Group: 18 TO <61 YEARS | A/H3N2C Age Group: 18 TO <61 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥61 YEARS | A/H3N2C + MF59 Age Group: ≥61 YEARS | A/H3N2C Age Group: ≥61 YEARS
Number analyzed (Participants) | 46 | 54 | 49 | 53 | 48 | 53 | 47 | 48 | 39 | 54 | 55 | 60
Percentages of Subjects
  Day 22 | 96 [85.2 to 99.5] | 98 [90.1 to 99.95] | 71 [56.7 to 83.4] | 89 [77 to 95.7] | 98 [88.9 to 99.95] | 85 [72.4 to 93.3] | 74 [59.7 to 86.1] | 90 [77.3 to 96.5] | 64 [47.2 to 78.8] | 57 [43.2 to 70.8] | 73 [59 to 83.9] | 63 [49.9 to 75.4]
  Day 43(N=43,53,48,52,49,53,46,46,39,53,55,59) | 100 [91.8 to 100] | 100 [93.3 to 100] | 92 [80 to 97.7] | 94 [84.1 to 98.8] | 98 [89.1 to 99.95] | 91 [79.3 to 96.9] | 85 [71.1 to 93.7] | 93 [82.1 to 98.6] | 67 [49.8 to 80.9] | 58 [44.1 to 71.9] | 80 [67 to 89.6] | 68 [54.4 to 79.4]

11. Secondary Outcome: Percentages of Subjects (3 to ≥ 61 Years of Age) Achieving HI Titers ≥1:40 Following Vaccination With H3N2 Monovalent Vaccine.
Description: The percentages of subjects achieving HI titers ≥1:40 against H3N2 homologous strain at three weeks after receiving first (day 22) and second (day 43) vaccination, is reported across age groups of 3 to ≥ 61 years.
Time Frame: Day 1, Day 22, Day 43 post vaccination
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- A/H3N2C + 1/2 MF59 Age Group: 18 TO <61 YEARS: Subjects 18 to <61years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75 µg antigen adjuvanted with half dose MF59.
- A/H3N2C Age Group: 18 TO <61 YEARS: Subjects 18 to <61years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
- A/H3N2C + 1/2 MF59 Age Group: ≥61 YEARS: Subjects ≥61 years old received two injections of cell-culture derived H3N2c vaccine, each dose containing 3.75µg antigen adjuvanted with half dose MF59.
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <61 YEARS | A/H3N2C + MF59 Age Group: 18 TO <61 YEARS | A/H3N2C Age Group: 18 TO <61 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥61 YEARS | A/H3N2C + MF59 Age Group: ≥61 YEARS | A/H3N2C Age Group: ≥61 YEARS
Number analyzed (Participants) | 52 | 55 | 50 | 54 | 51 | 53 | 48 | 49 | 39 | 55 | 56 | 61
Percentages of Subjects
  Day 1 | 8 [2.1 to 18.5] | 7 [2 to 17.6] | 14 [5.8 to 26.7] | 44 [30.9 to 58.6] | 59 [44.2 to 72.4] | 49 [35.1 to 63.2] | 60 [45.3 to 74.2] | 67 [52.5 to 80.1] | 74 [57.9 to 87] | 53 [38.8 to 66.3] | 54 [39.7 to 67] | 44 [31.5 to 57.6]
  Day 22(N=46,54,49,53,48,53,47,48,39,54,55,60) | 96 [85.2 to 99.5] | 98 [90.1 to 99.95] | 78 [63.4 to 88.2] | 100 [93.3 to 100] | 100 [92.6 to 100] | 98 [89.9 to 99.95] | 98 [88.7 to 99.95] | 100 [92.6 to 100] | 90 [75.8 to 97.1] | 93 [82.1 to 97.9] | 100 [93.5 to 100] | 93 [83.8 to 98.2]
  Day 43(N=43,53,48,52,49,53,46,46,39,53,55,59) | 100 [91.8 to 100] | 100 [93.3 to 100] | 96 [85.7 to 99.5] | 100 [93.2 to 100] | 100 [92.7 to 100] | 100 [93.3 to 100] | 98 [88.5 to 99.94] | 100 [92.3 to 100] | 100 [91 to 100] | 96 [87 to 99.54] | 100 [93.5 to 100] | 95 [85.9 to 98.9]

12. Primary Outcome: Percentages of Subjects (3 to ≥ 65 Years of Age) Achieving HI Titers ≥1:40 Following Vaccination With H3N2 Monovalent Vaccine.
Description: The percentages of subjects (3 to ≥ 65 years of age) achieving HI titers ≥1:40 against H3N2 homologous strain at baseline (Day 1) and three weeks after receiving first (Day 22) and second (Day 43) vaccination are reported.
Time Frame: Day 1, Day 22, Day 43 post vaccination
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥65 YEARS | A/H3N2C + MF59 Age Group: ≥65 YEARS | A/H3N2C Age Group: ≥65 YEARS
Number analyzed (Participants) | 53 | 55 | 50 | 53 | 51 | 53 | 53 | 55 | 48 | 50 | 50 | 52
Percentages of Subjects
  Day 1 | 8 [2.1 to 18.2] | 7 [2 to 17.6] | 14 [5.8 to 26.7] | 45 [31.6 to 59.6] | 59 [44.2 to 72.4] | 49 [35.1 to 63.2] | 57 [42.3 to 70.2] | 67 [53.3 to 79.3] | 67 [51.6 to 79.6] | 56 [41.3 to 70] | 52 [37.4 to 66.3] | 46 [32.2 to 60.5]
  Day 22 (N=47,54,49,52,48,53,52,54,48,49,49,51) | 96 [85.5 to 99.5] | 98 [90.1 to 99.95] | 78 [63.4 to 88.2] | 100 [93.2 to 100] | 100 [92.6 to 100] | 98 [89.9 to 99.95] | 96 [86.8 to 99.53] | 100 [93.4 to 100] | 88 [74.8 to 95.3] | 94 [83.1 to 98.7] | 100 [92.7 to 100] | 96 [86.5 to 99.52]
  Day 43 (N=43,53,48,52,49,53,51,52,48,48,49,50) | 100 [91.8 to 100] | 100 [93.3 to 100] | 96 [85.7 to 99.5] | 100 [93.2 to 100] | 100 [92.7 to 100] | 100 [93.3 to 100] | 96 [86.5 to 99.52] | 100 [93.2 to 100] | 98 [88.9 to 99.95] | 98 [88.9 to 99.95] | 100 [92.7 to 100] | 96 [86.3 to 99.51]

13. Secondary Outcome: GMR in Subjects (3 to ≥ 61 Years of Age) of Post-vaccination Versus Pre-vaccination HI Antibody Titers Following Vaccination With H3N2 Monovalent Vaccine.
Description: GMR of post-vaccination versus pre-vaccination HI GMTs following vaccination with H3N2 monovalent vaccine is reported across subjects with age groups 3 to ≥ 61 years.
Time Frame: Day 22/Day 1, Day 43/Day 1, Day183/ Day 1, Day 366/Day 1
Population: Analysis was done on Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <61 YEARS | A/H3N2C + MF59 Age Group: 18 TO <61 YEARS | A/H3N2C Age Group: 18 TO <61 YEARS | A/H3N2C + 1/2 MF59 Age Group: ≥61 YEARS | A/H3N2C + MF59 Age Group: ≥61 YEARS | A/H3N2C Age Group: ≥61 YEARS
Number analyzed (Participants) | 46 | 54 | 49 | 53 | 50 | 53 | 47 | 48 | 39 | 54 | 55 | 60
Ratios
  Day22/Day1(N=46,54,49,53,48,53,47,48,39,54,55,60) | 22 [15 to 32] | 33 [23 to 47] | 11 [7.50 to 16] | 14 [9.76 to 19] | 15 [10 to 22] | 13 [8.91 to 18] | 7.8 [5.48 to 11] | 12 [8.62 to 17] | 4.93 [3.35 to 7.25] | 4.05 [2.93 to 5.59] | 6.73 [4.88 to 9.28] | 5.53 [4.07 to 7.52]
  Day43/Day1(N=43,53,48,52,49,53,46,46,39,53,55,59) | 59 [43 to 81] | 82 [62 to 109] | 23 [17 to 31] | 18 [13 to 25] | 21 [15 to 30] | 14 [10 to 20] | 7.1 [5.21 to 9.69] | 10 [7.61 to 14] | 6.04 [4.32 to 8.45] | 4.14 [3.07 to 5.56] | 6.57 [4.90 to 8.80] | 6.2 [4.68 to 8.22]
  Day183/ Day1,N=38,44,42,48,50,47,40,44,37,52,54,58 | 9.96 [7.25 to 14] | 17 [13 to 23] | 7.18 [5.32 to 9.70] | 6.76 [5.02 to 9.10] | 8.19 [6.12 to 11] | 6.38 [4.72 to 8.62] | 3.98 [2.87 to 5.51] | 5.23 [3.86 to 7.09] | 4.30 [3.08 to 6.00] | 2.69 [2.03 to 3.55] | 3.82 [2.90 to 5.03] | 3.56 [2.73 to 4.65]
  Day 366/Day1,N=37,43,38,48,50,47,38,41,37,53,52,58 | 4.55 [3.22 to 6.42] | 8.26 [6.02 to 11] | 4.09 [2.91 to 5.75] | 4.43 [3.20 to 6.14] | 4.20 [3.06 to 5.78] | 4.15 [2.98 to 5.77] | 2.73 [2.00 to 3.73] | 4.21 [3.13 to 5.67] | 3.03 [2.22 to 4.14] | 1.69 [1.32 to 2.18] | 2.35 [1.82 to 3.04] | 2.37 [1.86 to 3.01]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 366.
Description: All solicited AEs and unsolicited AEs were collected from Day 1 to Day 7; any unsolicited AEs, any SAEs, medically attended AEs, AEs leading to withdrawal from the study, AESI and NOCD were collected from Day 1 (from 30 minutes) to Day 366 after every vaccination.
  Analysis was done on the safety data sets.
Groups:
- A/H3N2C Age Group: >=65 YEARS: Subjects ≥65 years old received two injections of a non-adjuvanted cell-culture derived H3N2c vaccine, each dose containing 15 µg antigen.
Arm/Group | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS | A/H3N2C Age Group: 3 TO <9 YEARS | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS | A/H3N2C Age Group: 9 TO <18 YEARS | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS | A/H3N2C Age Group: 18 TO <65 YEARS | A/H3N2C + 1/2 MF59 Age Group: >=65 YEARS | A/H3N2C + MF59 Age Group: >=65 YEARS | A/H3N2C Age Group: >=65 YEARS
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/54 | 0/50 | 0/54 | 0/51 | 1/53 | 3/51 | 0/54 | 1/48 | 2/52 | 5/49 | 5/51
Other Adverse Events (participants affected / at risk) | 36/50 | 46/54 | 30/50 | 44/54 | 42/51 | 45/53 | 35/51 | 43/54 | 30/48 | 33/52 | 31/49 | 32/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS (N=50) | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS (N=54) | A/H3N2C Age Group: 3 TO <9 YEARS (N=50) | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS (N=54) | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS (N=51) | A/H3N2C Age Group: 9 TO <18 YEARS (N=53) | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS (N=51) | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS (N=54) | A/H3N2C Age Group: 18 TO <65 YEARS (N=48) | A/H3N2C + 1/2 MF59 Age Group: >=65 YEARS (N=52) | A/H3N2C + MF59 Age Group: >=65 YEARS (N=49) | A/H3N2C Age Group: >=65 YEARS (N=51)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SURGICAL FAILURE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
AORTIC RUPTURE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A/H3N2C + 1/2 MF59 Age Group: 3 TO <9 YEARS (N=50) | A/H3N2C + MF59 Age Group: 3 TO <9 YEARS (N=54) | A/H3N2C Age Group: 3 TO <9 YEARS (N=50) | A/H3N2C + 1/2 MF59 Age Group: 9 TO <18 YEARS (N=54) | A/H3N2C + MF59 Age Group: 9 TO <18 YEARS (N=51) | A/H3N2C Age Group: 9 TO <18 YEARS (N=53) | A/H3N2C + 1/2 MF59 Age Group: 18 TO <65 YEARS (N=51) | A/H3N2C + MF59 Age Group: 18 TO <65 YEARS (N=54) | A/H3N2C Age Group: 18 TO <65 YEARS (N=48) | A/H3N2C + 1/2 MF59 Age Group: >=65 YEARS (N=52) | A/H3N2C + MF59 Age Group: >=65 YEARS (N=49) | A/H3N2C Age Group: >=65 YEARS (N=51)
DIARRHOEA (Gastrointestinal disorders) | 1 | 5 | 1 | 5 | 5 | 6 | 8 | 15 | 4 | 7 | 4 | 5
NAUSEA (Gastrointestinal disorders) | 6 | 5 | 1 | 12 | 11 | 10 | 5 | 11 | 5 | 6 | 6 | 5
VOMITING (Gastrointestinal disorders) | 4 | 4 | 3 | 4 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 2
FATIGUE (General disorders) | 7 | 11 | 7 | 18 | 21 | 19 | 12 | 18 | 11 | 11 | 13 | 7
INJECTION SITE BRUISING (General disorders) | 0 | 2 | 3 | 0 | 2 | 1 | 0 | 1 | 2 | 2 | 0 | 3
INJECTION SITE ERYTHEMA (General disorders) | 4 | 5 | 1 | 1 | 4 | 2 | 0 | 7 | 1 | 4 | 3 | 4
INJECTION SITE HAEMORRHAGE (General disorders) | 3 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 1
INJECTION SITE INDURATION (General disorders) | 4 | 7 | 0 | 3 | 9 | 3 | 1 | 9 | 1 | 2 | 2 | 3
INJECTION SITE PAIN (General disorders) | 31 | 38 | 23 | 39 | 37 | 33 | 26 | 35 | 22 | 15 | 23 | 7
MALAISE (General disorders) | 9 | 11 | 3 | 13 | 15 | 11 | 13 | 19 | 6 | 9 | 6 | 3
PYREXIA (General disorders) | 3 | 5 | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 2 | 4 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 | 5 | 2 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 3 | 2 | 10 | 12 | 7 | 4 | 7 | 4 | 8 | 3 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 5 | 5 | 10 | 6 | 9 | 8 | 7 | 5 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 | 3 | 2 | 10 | 10 | 6 | 8 | 11 | 9 | 5 | 6 | 5
HEADACHE (Nervous system disorders) | 8 | 7 | 4 | 19 | 19 | 15 | 15 | 18 | 13 | 9 | 8 | 6
SOMNOLENCE (Nervous system disorders) | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EATING DISORDER (Psychiatric disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IRRITABILITY (Psychiatric disorders) | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 4 | 0 | 0 | 0 | 1 | 2
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other